CLINICAL TRIAL: NCT03197064
Title: Effect of Fosaprepitant on Motor Evoked and Somatosensory Evoked Potentials Under General Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Mark Burbridge, Clinical Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-41444
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Results first posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Postoperative Nausea
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — fosaprepitant

STUDY DESIGN:
Intervention Model Description: A single group of up to 50 patients will be administered a standard dose of fosaprepitant 150 mg IV after induction of anesthesia. A standard neuromonitoring setup utilizing motor evoked potentials, and somatosensory evoked potentials will be used as indicated for the type of surgery. After baseline neuromonitoring measurements have been made, but prior to surgery starting, we will administer the fosaprepitant to determine if there are any effects on the motor evoked potentials or somatosensory evoked potentials measurements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Fosaprepitant (Other): Patients included in this study will be administered fosaprepitant 150 mg IV.
  Interventions: Drug: Fosaprepitant 150 mg

INTERVENTIONS:
Drug: Fosaprepitant 150 mg — Antiemetic used to prevent nausea and vomiting after general anesthesia.

SUMMARY:
The purpose of this study is to determine if intravenous fosaprepitant can interfere with nervous system monitoring signals in patients having surgery under general anesthesia. This medication has numerous effects on the sensory nerve transmission which can theoretically have effects on the ability to accurately measure somatosensory evoked potentials.

DETAILED DESCRIPTION:
The purpose of this study is to determine if intravenous fosaprepitant can interfere with nervous system monitoring signals in patients having surgery under general anesthesia. Fosaprepitant is a drug commonly used to prevent post-operative nausea and vomiting, and works by inhibiting "substance P", which is found in the brain and spinal cord. Theoretically, fosaprepitant could interfere with nervous system recordings because of its effect on substance P,but it is not known if this actually occurs. The drug will be given after the patient has been anesthetized but before surgical incision so that if there are any changes on the intraoperative neuromonitoring signals they can only be attributed to fosaprepitant.

If fosaprepitant alters intraoperative neuromonitoring signals during surgical procedures under general anesthesia, it would be important because anesthesiologist's who administer this drug would want to give it at the beginning of surgery when changes in intraoperative neuromonitoring signals would be unlikely to mean that these changes were due to surgical damage to the nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Having a surgical procedure requiring general anesthesia, having a surgical procedure where neuromonitoing with somatosensory evoked potentials and motor evoked potentials neuromonitoring is requested by the surgical team

Exclusion Criteria:

* Patient refusal, allergy to the drug or any of its excipients, pre-operative motor or sensory deficit

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Burbridge, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD available only to members of the research team involved in this project. All patient identifying information will be removed from all data as it is collected to protect patient privacy.

RESULTS

PARTICIPANT FLOW:
Groups:
- Fosaprepitant: Patients receive fosaprepitant 150 mg intravenously (i.v.).
Period: Overall Study
Arm/Group | Fosaprepitant
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fosaprepitant
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Somatosensory Evoked Potentials (SEPs), Extremity Amplitude (Left Upper Extremity)
Description: Neuromonitoring modality utilized during surgical procedures potentially affecting sensory component of central and peripheral nervous system.
  SEPs are the electrical signals generated by the nervous system in response to somatosensory stimuli - typically through electrical stimulation of the median nerve. SEPs are read on the skull with electroencephalography (EEG). SEPs was recorded using a 4-channel EEG system at baseline (predose) and regularly after study drug administration.
Time Frame: Baseline (pre-dose) and 30, 60, and 90 minutes post-dose
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Fosaprepitant
Number analyzed (Participants) | 11
µV
  Baseline | 2.685 (1.49)
  30 minutes | 2.545 (1.15)
  60 minutes | 2.58 (1.29)
  90 minutes | 2.292 (1.02)
Statistical Analysis 1: Comparison: Fosaprepitant; Difference in left upper extremity amplitude between baseline (pre-dose) and 30 minutes post-dose; Test type: Other; p = 0.35, t-test, 2 sided
Statistical Analysis 2: Comparison: Fosaprepitant; Difference in left upper extremity amplitude between baseline (pre-dose) and 60 minutes post-dose; Test type: Other; p = 0.47, t-test, 2 sided
Statistical Analysis 3: Comparison: Fosaprepitant; Difference in left upper extremity amplitude between baseline (pre-dose) and 90 minutes post-dose; Test type: Other; p = 0.066, t-test, 2 sided

2. Primary Outcome: Somatosensory Evoked Potentials (SEPs), Extremity Amplitude (Right Upper Extremity)
Description: as for outcome 1
Time Frame: Baseline (pre-dose) and 30, 60, and 90 minutes post-dose
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Fosaprepitant
Number analyzed (Participants) | 11
µV
  Baseline | 2.38 (1.35)
  30 minutes | 2.47 (1.05)
  60 minutes | 2.27 (1.01)
  90 minutes | 2.47 (1.2)
Statistical Analysis 1: Comparison: Fosaprepitant; Difference in right upper extremity amplitude between baseline (pre-dose) and 30 minutes post-dose; Test type: Other; p = 0.72, t-test, 2 sided
Statistical Analysis 2: Comparison: Fosaprepitant; Difference in right upper extremity amplitude between baseline (pre-dose) and 60 minutes post-dose; Test type: Other; p = 0.72, t-test, 2 sided
Statistical Analysis 3: Comparison: Fosaprepitant; Difference in right upper extremity amplitude between baseline (pre-dose) and 90 minutes post-dose; Test type: Other; p = 0.78, t-test, 2 sided

3. Primary Outcome: Somatosensory Evoked Potentials (SEPs), Extremity Amplitude (Left Lower Extremity)
Description: as for outcome 1
Time Frame: Baseline (pre-dose) and 30, 60, and 90 minutes post-dose
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Fosaprepitant
Number analyzed (Participants) | 11
µV
  Baseline | 1.56 (0.854)
  30 minutes | 1.56 (0.831)
  60 minutes | 1.47 (0.67)
  90 minutes | 1.35 (0.693)
Statistical Analysis 1: Comparison: Fosaprepitant; Difference in left lower extremity amplitude between baseline (pre-dose) and 30 minutes post-dose; Test type: Other; p = 0.93, t-test, 2 sided
Statistical Analysis 2: Comparison: Fosaprepitant; Difference in left lower extremity amplitude between baseline (pre-dose) and 60 minutes post-dose; Test type: Other; p = 0.39, t-test, 2 sided
Statistical Analysis 3: Comparison: Fosaprepitant; Difference in left lower extremity amplitude between baseline (pre-dose) and 90 minutes post-dose; Test type: Other; p = 0.08, t-test, 2 sided

4. Primary Outcome: Somatosensory Evoked Potentials (SEPs), Extremity Amplitude (Right Lower Extremity)
Description: as for outcome 1
Time Frame: Baseline (pre-dose) and 30, 60, and 90 minutes post-dose
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Fosaprepitant
Number analyzed (Participants) | 11
µV
  Baseline | 1.7 (0.911)
  30 minutes | 1.77 (1.09)
  60 minutes | 1.81 (1.08)
  90 minutes | 1.79 (1.18)
Statistical Analysis 1: Comparison: Fosaprepitant; Difference in right lower extremity amplitude between baseline (pre-dose) and 30 minutes post-dose; Test type: Other; p = 0.42, t-test, 2 sided
Statistical Analysis 2: Comparison: Fosaprepitant; Difference in right lower extremity amplitude between baseline (pre-dose) and 60 minutes post-dose; Test type: Other; p = 0.37, t-test, 2 sided
Statistical Analysis 3: Comparison: Fosaprepitant; Difference in right lower extremity amplitude between baseline (pre-dose) and 90 minutes post-dose; Test type: Other; p = 0.49, t-test, 2 sided

5. Primary Outcome: Motor Evoked Potentials Amplitude (Left Upper Extremity)
Description: Neuromonitoring modality utilized during surgical procedures affecting motor component of central and peripheral nervous system.
  MEPs are generated when stimulation of the brain on the motor cortex (with Transcranial Magnetic Stimulation [TMS]) causes the spinal cord and peripheral muscles to produce neuroelectrical signals. MEPs are typically measured in the hand muscles.
Time Frame: Baseline (pre-dose) and 30, 60, and 90 minutes post-dose
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Fosaprepitant
Number analyzed (Participants) | 11
µV
  Baseline | 1300 (1128.48)
  30 minutes | 1573.33 (1508.37)
  60 minutes | 1634.89 (1460.48)
  90 minutes | 1544.78 (1579.12)
Statistical Analysis 1: Comparison: Fosaprepitant; Difference in left upper extremity amplitude between baseline (pre-dose) and 30 minutes post-dose; Test type: Other; p = 0.386, t-test, 2 sided
Statistical Analysis 2: Comparison: Fosaprepitant; Difference in left upper extremity amplitude between baseline (pre-dose) and 60 minutes post-dose; Test type: Other; p = 0.388, t-test, 2 sided
Statistical Analysis 3: Comparison: Fosaprepitant; Difference in left upper extremity amplitude between baseline (pre-dose) and 90 minutes post-dose; Test type: Other; p = 0.247, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 6 hours
Arm/Group | Fosaprepitant
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT03197064/Prot_000.pdf